CLINICAL TRIAL: NCT05105360
Title: Prevention of Petersen's Hernia After Laparoscopic Gastrectomy for Gastric Cancer, Prospective, Multicenter Trial
Brief Title: Prevention of Petersen's Hernia After Laparoscopic Gastrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mefix study
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Petersen's Hernia

STUDY DESIGN:
Intervention Model Description: non-inferior study, multicenter, prospective, randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Petersen's closure group (Active Comparator): Petersen's space closure method
  Interventions: Procedure: Closure method of Petersen's space
- Mefix group (Experimental): Mesentery fixation method
  Interventions: Procedure: Mesentery fixation method

INTERVENTIONS:
Procedure: Closure method of Petersen's space — Surgeons closed Petersen's space between the mesentery of the jejunal Roux limb and the mesentery of the transverse colon at the posterior side of esophago-jejunostomy or gastro-jejunostomy from the mesentery root to the bowel side using a nonabsorbable barbed suture V-LocTM 3-0 (Medtronic VR, Minneapolis, MN, USA).
  Arms: Petersen's closure group
Procedure: Mesentery fixation method — Surgeons fixed the jejunal mesentery (jejunojejunostomy[J-J] distal 30 cm) to the transverse mesocolon using non-absorbable barbed suture VLocTM 3-0 sutures. The suture area was exposed by grasping the jejunum side mesentery (jejunal side, at site 30cm distal J-J) and the transverse mesocolon (colonic side). The jejunal side mesentery was fixed to the colonic side mesocolon between the jejunum and the transverse colon using nonabsorbable barbed V-LocTM 3-0 sutures.The suture started between jejunal mesentery just below of SMA vascular arcade and transverse mesocolon, and it finished when it reaches the root of the mesentery. To anchor the mesentery, continuous suturing with V-Loc two-point backward sutures were performed at the final step.
  Arms: Mefix group

SUMMARY:
* Aim of this study To compare the cases underwent operation to treat intestinal obstruction caused by Peterson hernia within 3 years after laparoscopic gastrectomy between closure method and Mefix methods.
* Primary end point: The cases underwent operation to treat intestinal obstruction caused by Peterson hernia within 3 years after laparoscopic gastrectomy was not- inferior between Closure and MEFIX.
* Secondary endpoint: Procedures' times (minutes), bleeding, Hospital stays (days) Occurrence of postoperative small bowel obstruction within 30 days after surgery, Short-term complications within 30 days after surgery, Occurrence of Petersen's Hernia according to the use of anti-adhesion agents, anastomotic methods, CLOSURE or MEFIX previous surgical suture condition, hernia degree, and bowel condition (strangulation, perforation) at the timing of emergent operation for treatment of Petersen's Hernia obstructions

DETAILED DESCRIPTION:
1. Background

1. Petersen's hernia after gastrectomy Petersen's hernia was reported in 1900 by German surgeon Walther Petersen following the occurrence of an internal hernia after gastrectomy and gastrojejunostomy (G-J) 1[]. Petersen's hernia occurs in the free space posterior to a G-J site after any type of G-J and is caused by herniation of the small bowel through the defect between the small bowel mesentery and the transverse mesocolon.

   As shown in CT figure in Figure 1, the small bowel mesentery rotates and twists, leading to an emergency situation in which necrosis of the entire small intestine occurs due to decreased blood circulation of the small intestine The occurrence rate of Petersen's hernias after laparoscopic Roux-en-Y G-J is approximately 1.7~9.7%

   - Peterson's hernia can occur in the RNY esophagojejunal anastomosis after gastrectomy, or after the RNY gastrojejunostomy and Billroth type 2 anastomosis after distal gastrectomy. Also, it can occur after the obesity surgery RNY gastric bypass surgery.
2. The incidence of internal hernia has been reported to be higher in laparoscopic approaches than in open gastrectomy One possible cause of the increasing incidence of Petersen's hernias is the recent development of minimally invasive surgery. A higher incidence of internal hernia is reported in minimally invasive gastrectomy than in open gastrectomy.

   After open surgery, adhesion was made between the small bowel and the operative wound site, however with minimally invasive surgery, adhesion is remarkably decreased, not only because of the disappearance of the open wound in the upper abdomen but also the use of antiadhesive agent Therefore, non-absorbable sutures require the closure of Peterson's spaces, and according to report of Blockhuys M, the frequency of internal hernia decreased after closure of Petersen's space.

   The frequency of internal hernia significantly decreases when Peterson space closure is implemented compared to the group that performed mesentery defect closure only.
3. The problem of Petersen's space closure procedure The closure of the defect at Petersen's space can induce bleeding by injuring the mesenteric vessels, as well as small bowel ischemia, caused by injuring the peripheral mesenteric vessels near the small bowel lumen. It has also been reported that early postoperative obstruction could be due to jejunal kinking of the closing site of the mesenteric defect. The closure of mesenteric defects increased the risk for severe postoperative complications in the early postoperative phase (<30 days) following the closure, mainly because of kinking of the jejunostomy site. We also encountered kinking of the jejunojejunostomy in the early postoperative periods after gastrectomy. However, it is not easy to determine if the complications are because of kinking of the entero-entero anastomosis or the adhesion effect from the closure of Petersen's space. Peterson space closure is necessary, but it is difficult by technical problem to develop an easy method.
4. Previous study We conducted jejunal mesentery fixing (Mefix) to the transverse mesocolon with a non-absorbable suture to prevent of a Petersen's hernia.

The theory of the Mefix method is as follows. When the mesentery of the small intestine is fixed to the transverse mesocolon between the small bowel and the colon mesentery, the defect still remains. However, the small bowel does not enter the defect because the small bowel mesentery is fixed at the transverse mesocolon; consequently, a Petersen's hernia does not occur.

MEFIX method allowed partial herniation of bowel, but it prevent of total herniation. This prevent bowel infarction

We closed Petersen's space defect between March 1st, 2016 and Dec 31th, 2017 (N=49), and we performed the Mefix procedure between July 1st, 2017 and June 30th, 2018 (N=26). We classified patients into the Petersen's space closure group (closure group) and the mesentery fixing group (Mefix group). All patients visited the hospital at six months and one year after surgery, and a CT scan was performed to check for the recurrence of gastric cancer. We determined the incidence of Petersen's hernia by abdominal CT scan, and we found no incidence of Petersen's hernias in either group. The procedure times for mesentery fixing (3.7 ± 1.1 minutes) were significantly shorter than those for Petersen's space closures (7.5 ± 1.5 minutes) (p<0.001). However, a retrospective study and a small group of patients seem to require a large, prospective random study.

ELIGIBILITY:
Inclusion Criteria:

: histological proven primary gastric adenocarcinoma

* no evidence of other distant metastasis
* R0 resection
* laparoscopic or robotic gastrectomy
* and reconstructed by Roux-en-Y reconstruction or the Billroth II procedure
* patient with appropriate conditions of activity; 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
* patient who have not previously received chemotherapy or radiation treatment in the abdomen.
* patinet who signed the consent form
* cTNM stage I or II or III

Exclusion Criteria:

* active double cancer (synchronous and metachronous double cancer within 5 disease-free years),

  * carcinoma in situ,
  * open gastrectomy,
  * reconstructed by Billroth I procedure,
  * gastric cancer recurrence, ;a history of gastrectomy. ;
  * a patient who has the history of abdominal surgery except laparoscopic appendectomy and gallbladder resection, and laparoscopic gynecologic surgery due to benign disease, and Cesarean section.
  * a patient who need co-ordination for other organs in preoperative examination (However, laparoscopic cholecystectomy is included in the selection criteria due to gallbladder polyps, and gallbladder disease).
  * Pregnant women, lactating women
  * a patient with mental illness (a person diagnosed with mental illness in medical records)
  * a patient who are taking corticosteroid whole-body (including herbal medicine)
  * a patient who has an uncontrolled history of angina or myocardial infarction within six months of the study;
  * uncontrolled hypertension
  * a patient who has a serious respiratory disease that requires continuous oxygen therapy;

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2029-01-26 (Estimated)

PRIMARY OUTCOMES:
post-operative 3-yr Petersen's hernia incidence | post-operative 3-yr
  Petersen's hernia incidence with operation for hernia reduction due to severe abdominal pain

SECONDARY OUTCOMES:
Postoperative morbidity and bowel obstruction incidence | complication within 30 days after surgery
  incidence of intestinal obstruction and complication
subgroup analysis of antiadhesive agent use | complication within 30 days after surgery
  subgroup analysis of incidence of intestinal obstruction by antiadhesive agent use
subgroup analysis of gastrectomy range and reconstruction method | complication within 30 days after surgery
  subgroup analysis of incidence of complication by gastrectomy range and reconstruction method
post-operative 5-yr Petersen's hernia incidence | post-operative 5-yr
  Petersen's hernia incidence with operation for hernia reduction due to severe abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Sangho Jeong, MD, Study Chair — Gyeongsang National University Hospital
Locations (1):
- Gyeongsang National University Hospital, Changwon, Gyeongsandnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No
The using of data is possible if the principle investigaster was accept of other researchers study plan.

REFERENCES:
- [Result] Min JS, Jeong SH, Park JH, Kim TH, Hong SC, Jung EJ, Ju YT, Jeong CY, Lee JK, Park M, Lee YJ. Prevention of Petersen's hernia using jejunal mesentery fixing (Mefix). Minim Invasive Ther Allied Technol. 2022 Apr;31(4):580-586. doi: 10.1080/13645706.2020.1848872. Epub 2020 Dec 3. PMID 33269633
- [Derived] Park JK, Kim DH, Jeon TY, Jeong SH, Kim TH, Min JS, Kim RB, Lee YJ, Park JH, Son YG, Yoon KY, Seo KW, Kim KH, Kim Y, Chae HD, Hwang SH, Lee SH, Chung JH, Kim HI, Park DJ, Kim KH, Seo SH, Oh SJ, Lee WY, In Choi C. Comparison between the mesenteric fixation method (MEFIX) and conventional methods at preventing the occurrence of Petersen's hernia: a study protocol for a multicenter randomized controlled trial. Trials. 2024 Jan 2;25(1):7. doi: 10.1186/s13063-023-07841-9. PMID 38167216